CLINICAL TRIAL: NCT04990856
Title: Tumor Blood Flow After Physical Exercise in Breast Cancer and Lymphoma Patients (Exetumor3 Study)
Brief Title: Exercise and Tumor Blood Flow in Lymphoma And Breast Cancer Patients (EXETUMOR 3)
Acronym: EXETUMOR3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Ilkka Heinonen, Adj. prof, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T06/024/21
Record Dates: First submitted 2021-06-03; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Tumor
Keywords: tumor; PET; exercise; blood flow
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Blood flow of the tumor experimented
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — Tumor blood flow after acute exercise

SUMMARY:
Recent pre-clinical studies strongly suggest that due to dysfunctional vasculature and blunted sympathetic constriction in the tumor, tumor blood flow is increased even by 200% compared to resting values. However, to the best of our knowledge these blood flow aspects have never been addressed clinically. Therefore, this research aims at investigating tumor blood flow response to exercise in human cancer patients. To address this goal, in total twenty (20) newly diagnosed breast cancer and eight (8) lymphoma patients will be recruited for the present acute exercise and tumor perfusion clinical trial. To study the effect of acute physical exercise on tumor blood flow and its heterogeneity, 30 minute bicycle exercise will be used to exercise these patients. Tumor blood flow will be measured by positron emission tomography at rest before and after the exercise. If the hypothesis of increased blood flow in response to exercise will be detected, this project has the potential to increase the basic physiological and mechanistic understanding of tumor microvasculature function in humans, which is also clinically highly relevant and can have long-lasting influences in the field in the future. Thus, the results from the project can be a breakthrough for cancer treatment, its mechanistic arguments, and thus renewal of evidence-based medicine and patient care.

DETAILED DESCRIPTION:
In regards to cancer, it would be reasonable to assume that also cancer behaves like all other inactive tissues in a body during exercise, meaning that also blood flow in the tumor environment is reduced particularly when exercise intensity increases. However, recent pre-clinical studies suggest that due to dysfunctional vasculature and blunted sympathetic constriction in the tumor, tumor blood flow is increased even by 200% compared to resting values (6; 18; 19) as increased cardiac output and blood pressure enhance perfusion pressure in the tumor. This improves its oxygenation (6; 18; 19), which is important as tumor hypoxia negatively affects the efficacy of treatment (27). Tumor hypoxia is promoted by heterogeneous blood flow in the tumor, but according to these pre-clinical studies exercise reduces the heterogeneity of tumor perfusion. However, it is not currently known if this is the case in patients, and it might be that tumor perfusion is actually decreased during exercise, but increased post-exercise, but this has never been addressed in clinical patients and is therefore the aim of the present study. Importantly, advanced imaging methods are available to investigate whether these pre-clinical findings can be extended to humans to serve as an evidence based proof-of-concept for the possible inclusion of exercise in the treatment of cancer during chemotherapy.

OBJECTIVES AND PURPOSE

The most important objective of this directly translatable and highly inter- disciplinary imaging, physical activity, health and medical research in the acute exercise study setting is:

To investigate whether acute moderate intensity exercise increases tumor blood flow

-It is hypothesized and expected that exercise increases tumor blood flow, documented as perfusion increase after acute exercise

STUDY DESIGN Each subject will serve their own control (tumor blood flow at rest vs. blood flow after exercise). Tumor blood flow will be measured with positron emission tomography (PET). To study the effect of acute physical exercise on tumor blood flow and its heterogeneity, bicycle exercise before PET scan will be used to exercise breast cancer and lymphoma cancer patients. These experiments are additional measurements to their normal treatments, and no new interventional approaches will be conducted in this study.

ELIGIBILITY:
Inclusion Criteria:

* a disease of newly diagnosed breast cancer, Hodgkin lymphoma, recurrent Hodgkin lymphoma and non-Hodgkin lymphoma with neck and thorax involvement.

Exclusion Criteria:

* abnormal fatigue, anemia, or physical dysfunction due to the disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-08-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood flow | up to 12 months
  Blood flow measured by PET imaging

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Heinonen, Principal Investigator — Turku PET Centre
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: up to 12 months